CLINICAL TRIAL: NCT05020405
Title: The Effect of Simvastatin With Guided Bone Regeneration on Ridge Volume in Ridge Splitting and Simultaneously Implantation: a Randomized Clinical Trial
Brief Title: The Effect of Simvastatin With Guided Bone Regeneration in Ridge Splitting and Simultaneously Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Dalia Rasheed Issa, principle investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200- 22
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Ridge Splitting; Simvastatin; Immediate Implant
MeSH Terms: interventions — 4-azido-2-nitrophenyluridylyl pyrophosphate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARS with GBR and SMV (Experimental): alveolar ridge splitting in combination with the use of GBR with SMV with immediate implant placement
  Interventions: Procedure: Immediate implant placement and ARS with GBR and SMV
- alveolar ridge splitting with GBR (Active Comparator): alveolar ridge splitting in combination with the use of GBR without SMV with immediate implant placement
  Interventions: Procedure: Immediate implant placement and ARS with GBR

INTERVENTIONS:
Procedure: Immediate implant placement and ARS with GBR and SMV — Implant insertion and GBR for augmentation of the gap between buccal and lingual plate using bone graft mixed with SMV
  Arms: ARS with GBR and SMV
Procedure: Immediate implant placement and ARS with GBR — Implant insertion and GBR for augmentation of the gap between buccal and lingual plate
  Arms: alveolar ridge splitting with GBR

SUMMARY:
Ridge split augmentation technique, with immediate implant placement, reduces the time of the treatment and the time of the final prosthetic reconstruction. Furthermore, compression of the bone increases its density. SMV is also found to promote osteogenic differentiation of bone marrow stem cells, suppress osteoclastic differentiation in bone tissue, and promotes osseointegration around implants in animal studies. The aim of this study is to compare surgical outcomes of the application of the alveolar ridge splitting (ARS) in combination with guided bone regeneration (GBR) using bone grafting and a barrier membrane, associated with immediate implant placement versus ARS in combination with the use of SMV with GBR using bone grafting and a barrier membrane, associated with immediate implant placement in patients with horizontally atrophic jaw bones.

ELIGIBILITY:
Inclusion Criteria:

* good general health at the time of surgery.
* at least 3 months of healing after tooth extraction.
* horizontally compromised alveolar ridges at least 10 mm high and 3 mm wide.

Exclusion Criteria:

* a vertical bone defect in the edentulous ridge.
* thick cortex in the labial/buccal with less cancellous bone inside
* obvious undercut on the labial/buccal side.
* uncontrolled periodontal conditions or other oral disorders.
* history of radiotherapy in the head and neck region.
* uncontrolled diabetes mellitus or other systematic disorders.
* smokers.
* Pregnancy.
* non-compliant patients.
* allergic reaction to the medications used.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Measurements of the amount of bone formation in millimeters around immediately placed dental implants | 9 months
  Measurements of the amount of bone formation in millimeters using GBR with or without the combined effect of SMV in the ridge splitting following immediate implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Dalia R Issa, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Faculty of Dentistry, Kafrelsheikh University, Kafr ash Shaykh, Egypt

REFERENCES:
- [Derived] Issa DR, Elamrousy W, Gamal AY. Alveolar ridge splitting and simvastatin loaded xenograft for guided bone regeneration and simultaneous implant placement: randomized controlled clinical trial. Clin Oral Investig. 2024 Jan 4;28(1):71. doi: 10.1007/s00784-023-05427-y. PMID 38172458